CLINICAL TRIAL: NCT06840483
Title: Phase 2 Study of Zelenectide Pevedotin in Participants With NECTIN4 Amplified Advanced Breast Cancer
Brief Title: Study of Zelenectide Pevedotin in Participants With Advanced Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BicycleTx Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BT8009-201 (Duravelo-3); 2024-517868-33-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-18; First posted 2025-02-21 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: NECTIN4; Zelenectide pevedotin; HR+/HER2-negative; TNBC; Chemotherapy; Duravelo-3; Advanced Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (HR+/HER2-negative breast cancer) (Experimental)
  Interventions: Drug: Zelenectide pevedotin (BT8009)
- Cohort B (TNBC) (Experimental)
  Interventions: Drug: Zelenectide pevedotin (BT8009)

INTERVENTIONS:
Drug: Zelenectide pevedotin (BT8009) — Participants will receive zelenectide pevedotin on Days 1, and 8 of every 21-day cycle.

SUMMARY:
This is a global, multicenter, open-label study that aims to assess the efficacy and safety of zelenectide pevedotin in participants with NECTIN4-amplified recurrent, unresectable, or metastatic breast cancer who have received prior therapy (see inclusion criteria below). The study will comprise of 2 cohorts. Cohort A will include participants with hormone receptor positive/ human epidermal growth factor receptor 2 negative [HR+/HER2-] breast cancer, whereas Cohort B will include participants with triple-negative breast cancer (TNBC).

ELIGIBILITY:
Inclusion Criteria

* Archival or fresh tumor tissue comprised of TNBC or HR+/HER2-negative invasive breast cancer available for NECTIN4 gene amplification testing.
* Confirmed NECTIN4 gene amplification by an analytically validated clinical trial assay (CTA).
* Measurable disease as defined by RECIST v1.1.
* Life expectancy ≥ 12 weeks.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of ≤ 1.

  1. Cohort A Specific Inclusion Criteria: Histologically or cytologically confirmed HR+/HER2-negative endocrine resistant/refractory breast cancer according to ASCO-CAP guidelines and received at least 1 and up to 3 prior lines of non-endocrine-based therapy for advanced disease.
  2. Cohort B Specific Inclusion Criteria: Histologically or cytologically confirmed TNBC, including ER-low positive breast cancers (1-10% of cells expressing hormonal receptors by IHC), according to ASCO-CAP guidelines and have received at least 1 and up to 3 prior lines of systemic therapy for advanced disease.

Exclusion Criteria

* Prior treatment with any antibody drug conjugate (ADC) containing an Monomethyl Auristatin E (MMAE) (vedotin) payload or other MMAE-based therapy.
* Known hypersensitivity or allergy to any of the ingredients of any of the study interventions, or to MMAE.
* Previously tested HER2-positive (IHC 3+ or ISH+) on prior pathology testing (per ASCO-CAP guidelines).
* Active keratitis or corneal ulcerations.
* Active or untreated central nervous system (CNS) metastases.
* Uncontrolled diabetes or hypertension.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently).
* Active interstitial lung disease or pneumonitis requiring ongoing treatment with steroids (>10mg/day of prednisone or equivalent) or other immunosuppressive medications.
* Requirement, while on study, for treatment with strong inhibitors or strong inducers of human cytochrome P450 3A (CYP3A) or inhibitors of P-glycoprotein (P-gp) including herbal- or food-based inhibitors.
* Prior treatment with any systemic anticancer therapy within 28 days or 5 half-lives, whichever is shorter, prior to first dose of study treatment

Note: Additional protocol defined Inclusion/Exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors per RECIST version 1.1 as assessed by the Investigator | Up to approximately 3 years
  Percentage of participants with either a confirmed complete response (CR) or partial response (PR)

SECONDARY OUTCOMES:
Number of participants reporting adverse events (AEs) and Serious adverse events (SAEs) | Up to approximately 3 years
  Safety and tolerability will be reported as incidence, severity, seriousness, relationship, and type of treatment-emergent adverse events, abnormalities in laboratory, electrocardiogram (ECG), vital signs and treatment modifications using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 criteria.
Duration of Response (DOR) per RECIST v1.1 as assessed by the Investigator | Up to approximately 3 years
  DoR as measured by the time from first documentation of objective response to the first documentation of disease progression assessed by the Investigator or to death (due to any cause), whichever occurs first.
Disease Control Rate (DCR) per RECIST v1.1 as assessed by the Investigator | Up to approximately 3 years
  Percentage of participants with confirmed CR, PR, or stable disease (SD)
Clinical Benefit Rate (CBR) per RECIST v1.1 as assessed by the Investigator | Up to approximately 3 years
  Percentage of participants with CR, PR or SD ≥16 weeks
Progression Free Survival (PFS) per RECIST v1.1 as assessed by the Investigator | Up to approximately 3 years
  PFS is measured by the time from the first day of study drug administration (Day 1) to the first documentation of disease progression per RECIST v1.1 as assessed by the Investigator, or to death (due to any cause), whichever occurs first.
Overall Survival | Up to approximately 4 years
  OS is defined as length of time from the first day of study drug administration (Day 1) to death (due to any cause).
Time To Progression (TTP) per RECIST v1.1 as assessed by the Investigator | Up to approximately 4 years
  TTP is defined as the time from first dose of study drug administration until first documentation of disease progression.

CONTACTS AND LOCATIONS:
Locations (39):
- United States (21):
  - City of Hope National Medical Center, Duarte, California
  - University of Colorado Denver, Aurora, Colorado
  - Yale New Haven Hospital - Yale Cancer Center, New Haven, Connecticut
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (SKCCC), Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Siteman Cancer Center, St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center - Main Campus, New York, New York
  - Duke Cancer Institute, Durham, North Carolina
  - Compass Oncology - Rose Quarter Cancer Center, Portland, Oregon
  - SCRI Oncology Partners, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - O'Quinn Medical Tower - McNair Campus (Baylor College of Medicine Medical Center), Houston, Texas
  - Texas Oncology San Antonio, San Antonio, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia
- Belgium (3):
  - Institut Jules Bordet, Brussels
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
- France (3):
  - Centre Leon Berard, Lyon
  - Centre de Lutte Contre le Cancer - Centre Eugene Marquis, Rennes
  - Oncopole Claudius Regaud, Toulouse
- Italy (4):
  - Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - IRCCS IRST, Meldola, Forli/Cesena
  - Clinica Oncologica-Azienda Ospedaliero Universitaria delle Marche, Ancona
  - Istituto Europeo di Oncologia, Milan
  - S.C. Oncologia Clinica Sperimentale di Senologia - IRCCS Fondazione Pascale, Napoli
- Spain (4):
  - Hospital Quironsalud Barcelona, Barcelona
  - Hospital Beata Maria Ana, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Centro Integral Oncologico Clara Campal, Madrid
- United Kingdom (3):
  - Barts Health NHS Trust, London
  - The Royal Marsden NHS Foundation Trust, London
  - The Royal Marsden NHS Foundation Trust, Sutton

IPD SHARING:
Plan to Share IPD: No